CLINICAL TRIAL: NCT01517477
Title: A Prospective, Randomized, Controlled Evaluation of Open-Angle Glaucoma Subjects on Two Topical Hypotensive Medications, Implanted With One, Two, or Three Trabecular Micro-Bypass Stents
Brief Title: One, Two, or Three iStents for the Reduction of Intraocular Pressure in Open-angle Glaucoma Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCF-033
Record Dates: First submitted 2012-01-23; First posted 2012-01-25 (Estimated); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Primary Open Angle Glaucoma (POAG)
Keywords: Open angle; Glaucoma; surgery; Glaucoma, Open-Angle; Ocular Hypertension; Eye Diseases
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Ocular Hypertension; Eye Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- First Arm: One iStent (Experimental): Device: One iStent
  Interventions: Device: iStent
- Second Arm: Two iStents (Experimental): Device: Two iStent devices
  Interventions: Device: iStent
- Third Arm: Three iStents (Experimental): Device: Three iStent devices
  Interventions: Device: iStent

INTERVENTIONS:
Device: iStent — Implantation of One iStent through a small temporal clear corneal incision.
  Arms: First Arm: One iStent
Device: iStent — Implantation of Two iStents through a small temporal clear corneal incision
  Arms: Second Arm: Two iStents
Device: iStent — Implantation of Three iStents through a small temporal clear corneal incision
  Arms: Third Arm: Three iStents

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the intraocular pressure (IOP) lowering effect of one, two, or three iStent devices in eyes of subjects previously on two anti-glaucoma medications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open-angle glaucoma (POAG)
* Subject on two topical hypotensive medications

Exclusion Criteria:

* Traumatic, uveitic, neovascular, or angle closure glaucoma
* Fellow eye already enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Mean diurnal intraocular pressure (IOP) reduction of greater than or equal to 20% at month 12 vs. baseline | 12 Months

SECONDARY OUTCOMES:
Mean diurnal IOP <18 mmHg at month 12 | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- S.V. Malayan's Ophthalmology Centre, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: Yes
18 month results published in Clinical Ophthalmology 2015:9 2313-2320.